CLINICAL TRIAL: NCT03351478
Title: A 26-week Randomized, Double-blind, Controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin Compared to Empagliflozin, and Placebo in Participants With Type 2 Diabetes Who Have Inadequate Glycemic Control on Dipeptidyl Peptidase 4 Inhibitor (DPP4(i)) With or Without Metformin
Brief Title: Efficacy and Safety of Sotagliflozin Versus Placebo and Empagliflozin in Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control While Taking a DPP4 Inhibitor Alone or With Metformin
Acronym: SOTA-EMPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC14867; 2016-001803-22 (EudraCT Number); U1111-1190-7607 (Other: UTN)
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sotagliflozin 400 mg (Experimental): Following a 2-week run-in period, sotagliflozin 400 mg (milligrams) administered as two 200 mg tablets and one placebo capsule (identical to the empagliflozin capsule in appearance), once daily before the first meal of the day for up to 26 weeks.
  Interventions: Drug: Sotagliflozin; Drug: Placebo
- Empagliflozin 25 mg (Active Comparator): Following a 2-week run-in period, placebo matching sotagliflozin administered as two tablets (identical to sotagliflozin in appearance) and one capsule of empagliflozin 25 mg, once daily before the first meal of the day for up to 26 weeks.
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Placebo (Placebo Comparator): Following a 2-week run-in period, placebo was given as two placebo tablets (identical to sotagliflozin) and one placebo capsule (identical to empagliflozin) once daily before the first meal of the day for up to 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin 400 mg was administered as two tablets, once daily before the first meal of the day.
  Other Names: SAR439954
  Arms: Sotagliflozin 400 mg
Drug: Empagliflozin — Empagliflozin 25 mg capsule was administered, once daily before the first meal of the day.
  Arms: Empagliflozin 25 mg
Drug: Placebo — Placebo was administered as two tablets (identical to sotagliflozin in appearance), once daily before the first meal of the day.
  Arms: Empagliflozin 25 mg; Placebo
Drug: Placebo — Placebo was administered as one capsule (identical to the empagliflozin capsule in appearance), once daily before the first meal of the day.
  Arms: Sotagliflozin 400 mg

SUMMARY:
The purpose of the study is to demonstrate the superiority of sotagliflozin versus placebo on hemoglobin A1c (HbA1c) reduction in participants with type 2 diabetes (T2D) who have inadequate glycemic control on a DPP4(i) with or without metformin.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes on Dipeptidyl peptidase-4 inhibitors(DPP4(i)) with or without metformin at a stable dose for at least 12 weeks prior to Screening Visit. Metformin dose will be ≥1500 mg per day (or maximum tolerated dose [documented]). DPP4(i) dose must be the appropriate dose as per local label.
* Signed written informed consent.

Exclusion criteria:

* Body mass index (BMI) ≤20 kg/m^2 or >45 kg/m^2 at Screening.
* Use of any antidiabetic drug other than DPP4 inhibitors and metformin within 12 weeks preceding the Screening Visit.
* Participants who have previously participated in any clinical trial of sotagliflozin/LX4211.
* Use of a selective sodium-glucose co-transporter type 2 (SGLT2) inhibitor (e.g., canagliflozin, dapagliflozin, or empagliflozin) within 3 months prior to the screening visit.
* Participants with severe anemia, severe cardiovascular disease (including congestive heart failure New York Heart Association IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease or participants with a short life expectancy that, according to Investigator, will preclude their safe participation in this study, or will make the implementation of the protocol or interpretation of the study results difficult.
* Current diagnosis of chronic hepatitis and/or other clinically active liver disease requiring treatment.
* Participants with contraindication to empagliflozin as per local labelling.
* Participants with contraindication to metformin as per local labelling.
* Hemoglobin A1c <7.0% or >11.0% at Screening (central laboratory).
* Fasting plasma glucose >270 mg/dL (>15.0 mmol/L) measured by the central laboratory at Screening (Visit 1), and confirmed by a repeat test (>270 mg/dL [>15.0 mmol/L]) before Randomization.
* Previous use of any type of insulin for >1 month (except for treatment of gestational diabetes).
* Pregnant (confirmed by serum pregnancy test at Screening) or breast-feeding women.
* Women of childbearing potential not willing to use highly effective method(s) of birth control during the study treatment period and follow-up period, or who are unwilling or unable to be tested for pregnancy during the study.
* Mean of 3 separate blood pressure (BP) measurements >180 mmHg (systolic blood pressure [SBP]) or >100 mmHg (diastolic blood pressure [DBP]).
* History of the hypertensive crisis resulting in emergency medical care within 12 weeks prior to Screening Visit.
* Lower extremity complications (such as skin ulcers, infection, osteomyelitis, and gangrene) identified during the Screening period, and still requiring treatment at Randomization.
* Laboratory findings with the central laboratory tests at Visit 1:
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of the normal laboratory range (ULN);
* Total bilirubin >1.5 times the ULN (except in case of Gilbert's syndrome);
* Neutrophils <1 500/mm^3 (or according to ethnic group) and/or platelets <100 000/mm^3;
* Amylase and/or lipase >3 times the ULN;
* Participants with renal impairment as defined by the estimated glomerular filtration rate (eGFR) criterion that precludes initiation of empagliflozin as per the approved local label (eg, <45 mL/min/1.73 m^2 in US; <60 mL/min/1.73 m^2 in EU).
* Secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
* If the participant is on hypertensive medications, the antihypertensive has been changed in the 8 weeks prior to Screening (new drug or new dose).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (160):
- United States (53):
  - Investigational Site Number 8408035, Birmingham, Alabama
  - Investigational Site Number 8408028, Sheffield, Alabama
  - Investigational Site Number 8408047, Hawaiian Gardens, California
  - Investigational Site Number 8408031, Spring Valley, California
  - Investigational Site Number 8408067, Van Nuys, California
  - Investigational Site Number 8408069, Northglenn, Colorado
  - Investigational Site Number 8408009, Miami, Florida
  - Investigational Site Number 8408049, Ocoee, Florida
  - Investigational Site Number 8408005, Orlando, Florida
  - Investigational Site Number 8408040, Orlando, Florida
  - Investigational Site Number 8408019, Palmetto Bay, Florida
  - Investigational Site Number 8408064, Port Charlotte, Florida
  - Investigational Site Number 8408061, Columbus, Georgia
  - Investigational Site Number 8408074, Macon, Georgia
  - Investigational Site Number 8408079, Savannah, Georgia
  - Investigational Site Number 8408059, Statesboro, Georgia
  - Investigational Site Number 8408051, Blackfoot, Idaho
  - Investigational Site Number 8408033, Elgin, Illinois
  - Investigational Site Number 8408003, New Orleans, Louisiana
  - Investigational Site Number 8408002, Rockville, Maryland
  - Investigational Site Number 8408044, Fall River, Massachusetts
  - Investigational Site Number 8408008, Flint, Michigan
  - Investigational Site Number 8408027, West Seneca, New York
  - Investigational Site Number 8408037, Fayetteville, North Carolina
  - Investigational Site Number 8408053, Greensboro, North Carolina
  - Investigational Site Number 8408012, Greensboro, North Carolina
  - Investigational Site Number 8408013, Salisbury, North Carolina
  - Investigational Site Number 8408045, Oklahoma City, Oklahoma
  - Investigational Site Number 8408068, Warwick, Rhode Island
  - Investigational Site Number 8408060, Fort Mill, South Carolina
  - Investigational Site Number 8408018, Jefferson City, Tennessee
  - Investigational Site Number 8408010, Knoxville, Tennessee
  - Investigational Site Number 8408038, Knoxville, Tennessee
  - Investigational Site Number 8408072, Brownsville, Texas
  - Investigational Site Number 8408056, Dallas, Texas
  - Investigational Site Number 8408082, Dallas, Texas
  - Investigational Site Number 8408052, Dallas, Texas
  - Investigational Site Number 8408001, Houston, Texas
  - Investigational Site Number 8408032, Houston, Texas
  - Investigational Site Number 8408016, Houston, Texas
  - Investigational Site Number 8408017, Houston, Texas
  - Investigational Site Number 8408036, Houston, Texas
  - Investigational Site Number 8408022, Houston, Texas
  - Investigational Site Number 8408029, Katy, Texas
  - Investigational Site Number 8408054, McAllen, Texas
  - Investigational Site Number 8408039, Mesquite, Texas
  - Investigational Site Number 8408042, Plano, Texas
  - Investigational Site Number 8408011, San Antonio, Texas
  - Investigational Site Number 8408041, Schertz, Texas
  - Investigational Site Number 8408007, Bountiful, Utah
  - Investigational Site Number 8408026, Holladay, Utah
  - Investigational Site Number 8408006, Burke, Virginia
  - Investigational Site Number 8408004, Manassas, Virginia
- Bulgaria (11):
  - Investigational Site Number 1008011, Gabrovo
  - Investigational Site Number 1008006, Plovdiv
  - Investigational Site Number 1008001, Plovdiv
  - Investigational Site Number 1008005, Rousse
  - Investigational Site Number 1008007, Rousse
  - Investigational Site Number 1008002, Smolyan
  - Investigational Site Number 1008008, Sofia
  - Investigational Site Number 1008012, Sofia
  - Investigational Site Number 1008003, Stara Zagora
  - Investigational Site Number 1008010, Stara Zagora
  - Investigational Site Number 1008004, Varna
- Canada (10):
  - Investigational Site Number 1248001, Brampton
  - Investigational Site Number 1248007, Burlington
  - Investigational Site Number 1248003, Newmarket
  - Investigational Site Number 1248010, Québec
  - Investigational Site Number 1248009, Sherbrooke
  - Investigational Site Number 1248002, Thornhill
  - Investigational Site Number 1248004, Toronto
  - Investigational Site Number 1248011, Toronto
  - Investigational Site Number 1248005, Vancouver
  - Investigational Site Number 1248008, Victoriaville
- Czechia (12):
  - Investigational Site Number 2038007, Brandys
  - Investigational Site Number 2038003, Havířov
  - Investigational Site Number 2038004, Krnov
  - Investigational Site Number 2038011, Ostrava
  - Investigational Site Number 2038006, Pardubice
  - Investigational Site Number 2038010, Pilsen
  - Investigational Site Number 2038009, Prague
  - Investigational Site Number 2038013, Prague
  - Investigational Site Number 2038002, Prague
  - Investigational Site Number 2038005, Prague
  - Investigational Site Number 2038008, Prague
  - Investigational Site Number 2038001, Praha 10 - Uhrineves
- France (7):
  - Investigational Site Number 2508005, Corbeil-Essonnes
  - Investigational Site Number 2508006, La Roche-sur-Yon
  - Investigational Site Number 2508007, La Tronche
  - Investigational Site Number 2508003, Mulhouse
  - Investigational Site Number 2508002, Nantes
  - Investigational Site Number 2508001, Paris
  - Investigational Site Number 2508004, Saint-Mandé
- Italy (11):
  - Investigational Site Number 3808010, Catania
  - Investigational Site Number 3808003, Catania
  - Investigational Site Number 3808002, Chieti
  - Investigational Site Number 3808004, Milan
  - Investigational Site Number 3808005, Milan
  - Investigational Site Number 3808009, Pavia
  - Investigational Site Number 3808008, Roma
  - Investigational Site Number 3808001, Roma
  - Investigational Site Number 3808007, Roma
  - Investigational Site Number 3808011, San Giovanni Rotondo
  - Investigational Site Number 3808006, Siena
- Latvia (8):
  - Investigational Site Number 4288004, Kuldīga
  - Investigational Site Number 4288008, Limbaži
  - Investigational Site Number 4288003, Ogre
  - Investigational Site Number 4288007, Riga
  - Investigational Site Number 4288001, Riga
  - Investigational Site Number 4288002, Riga
  - Investigational Site Number 4288006, Sigulda
  - Investigational Site Number 4288005, Talsi
- Mexico (7):
  - Investigational Site Number 4848002, Chihuahua City
  - Investigational Site Number 4848003, Cuernavaca
  - Investigational Site Number 4848007, Durango, Durango
  - Investigational Site Number 4848011, Mexico City
  - Investigational Site Number 4848005, Monterrey
  - Investigational Site Number 4848001, Monterrey
  - Investigational Site Number 4848012, Monterrey
- Russia (14):
  - Investigational Site Number 6438008, Chelyabinsk
  - Investigational Site Number 6438006, Dzerzhinsky
  - Investigational Site Number 6438009, Kemerovo
  - Investigational Site Number 6438010, Novosibirsk
  - Investigational Site Number 6438013, Saint Petersburg
  - Investigational Site Number 6438003, Saint Petersburg
  - Investigational Site Number 6438014, Saint Petersburg
  - Investigational Site Number 6438002, Saint Petersburg
  - Investigational Site Number 6438005, Saint Petersburg
  - Investigational Site Number 6438001, Saint Petersburg
  - Investigational Site Number 6438012, Saratov
  - Investigational Site Number 6438015, Volgograd
  - Investigational Site Number 6438007, Vsevolozhsk
  - Investigational Site Number 6438011, Yaroslavl
- Slovakia (9):
  - Investigational Site Number 7038005, Bardejov
  - Investigational Site Number 7038009, Bratislava
  - Investigational Site Number 7038001, Košice
  - Investigational Site Number 7038006, Lučenec
  - Investigational Site Number 7038008, Nové Zámky
  - Investigational Site Number 7038004, Považská Bystrica
  - Investigational Site Number 7038002, Rožňava
  - Investigational Site Number 7038007, Sabinov
  - Investigational Site Number 7038003, Vrútky
- Spain (10):
  - Investigational Site Number 7248006, Barcelona
  - Investigational Site Number 7248002, Córdoba
  - Investigational Site Number 7248005, Malaga Malaga
  - Investigational Site Number 7248010, Santa Coloma de Gramenet
  - Investigational Site Number 7248009, Santiago de Compostela
  - Investigational Site Number 7248004, Seville
  - Investigational Site Number 7248008, Seville
  - Investigational Site Number 7248001, Seville
  - Investigational Site Number 7248003, Valencia
  - Investigational Site Number 7248007, Zaragoza
- United Kingdom (8):
  - Investigational Site Number 8268008, Darlington
  - Investigational Site Number 8268004, Dundee
  - Investigational Site Number 8268006, Exeter
  - Investigational Site Number 8268001, Hull
  - Investigational Site Number 8268002, Huntingdon
  - Investigational Site Number 8268007, Sheffield
  - Investigational Site Number 8268003, Southampton
  - Investigational Site Number 8268005, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) and supporting clinical documents are available for request at clinicalstudydatarequest.com. While making information available Sanofi continues to protect the privacy of the participants in clinical trials and to remove commercially confidential information (CCI). Details on Data Sharing criteria and process for requesting access can be found at this web address: clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 160 investigative sites in Bulgaria, Canada, Czechia, France, Italy, Latvia, Mexico, Russian Federation, Slovakia, Spain, United Kingdom, and the United States from 27 November 2017 to 16 May 2019.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were enrolled in 1 of 3 treatment groups, Sotagliflozin, Empagliflozin, or Placebo. Participants were randomly assigned in the ratio of 2:2:1 to these reporting groups.
Groups:
- Sotagliflozin 400 mg: Following a 2-week run-in period, sotagliflozin 400 milligrams (mg) administered as two 200 mg tablets and one placebo capsule (identical to empagliflozin capsule in appearance), once daily before the first meal of the day for up to 26 weeks.
- Placebo: Following a 2-week run-in period, placebo given as two placebo tablets (identical to sotagliflozin) and one placebo capsule (identical to empagliflozin) once daily before the first meal of the day for up to 26 weeks.
Period: Overall Study
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Started | 307 | 309 | 154
Completed | 293 | 292 | 147
Not Completed | 14 | 17 | 7
Not completed — At the subject's own request | 11 | 12 | 5
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Poor compliance to protocol | 1 | 0 | 0
Not completed — Reason not Specified | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Sotagliflozin 400 mg: Following a 2-week run-in period, sotagliflozin 400 mg administered as two 200 mg tablets and one placebo capsule (identical to empagliflozin capsule in appearance), once daily before the first meal of the day for up to 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo | Total
Number analyzed (Participants) | 307 | 309 | 154 | 770
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.7) | 59.7 (9.6) | 59.8 (9.6) | 59.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 158 | 75 | 374
  Male | 166 | 151 | 79 | 396
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 66 | 33 | 155
  Not Hispanic or Latino | 251 | 243 | 121 | 615
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 21 | 8 | 47
  Asian | 17 | 11 | 4 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 13 | 13 | 5 | 31
  White | 256 | 257 | 137 | 650
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 6 | 0 | 7
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.23 (0.84) | 8.21 (0.93) | 8.21 (0.93) | 8.22 (0.90)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 134.55 (13.56) | 131.64 (12.18) | 133.19 (12.53) | 133.11 (12.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) % at Week 26
Description: An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline, Week 26
Population: Intent-to-treat (ITT) population included all randomized participants. Missing data was imputed using the retrieved dropouts imputation method.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
percentage of HbA1c | -0.7 (0.1) | -0.8 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The change from baseline to Week 26 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and the country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Square (LS) Means = -0.43, 95% CI 2-sided [-0.62 to -0.25], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Empagliflozin 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.145, ANCOVA; Difference in LS Means = 0.12, 95% CI 2-sided [-0.04 to 0.28], Standard Error of Mean 0.08

2. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 12 in Participants With Baseline SBP ≥ 130 mmHg
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 12
Population: Participants from the ITT population, all randomized participants with data available at the given time point for analysis. Missing data was imputed using washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 146 | 151 | 84
mmHg | -5.6 (1.3) | -6.7 (1.3) | -3.5 (1.5)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The change from baseline to Week 12 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤ 8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No) and the country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.1529, ANCOVA; Difference in LS Means = -2.05, 95% CI 2-sided [-4.87 to 0.76], Standard Error of Mean 1.43
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Empagliflozin 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3377, ANCOVA; Difference in LS Means = 1.17, 95% CI 2-sided [-1.21 to 3.55], Standard Error of Mean 1.21

3. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose (PPG) Following a Mixed Meal at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 26
Population: ITT population included all randomized participants. Missing data was imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
millimole per liter (mmol/L) | -1.3 (0.2) | -1.2 (0.9) | -0.4 (0.2)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The change from baseline to Week 26 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and the country as fixed effects, and baseline 2-hour postprandial glucose as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -0.91, 95% CI 2-sided [-1.33 to -0.5], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Empagliflozin 25 mg; The change from baseline to Week 26 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), randomization strata of mean SBP (<130, ≥ 130 mmHg) at screening, and the country as fixed effects, and baseline 2-hour postprandial glucose as a covariate; Test type: Superiority; p = 0.8397, ANCOVA; Difference in LS Means = -0.03, 95% CI 2-sided [-0.37 to 0.3], Standard Error of Mean 0.17

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 26
Population: ITT population included all randomized participants. Missing data was imputed using the retrieved dropouts imputation method.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
mmol/L | -1.3 (0.2) | -1.6 (0.2) | -0.5 (0.2)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The change from baseline to Week 26 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and the country as fixed effects, and baseline fasting plasma glucose as a covariate; Test type: Superiority; p = 0.0005, ANCOVA; Difference in LS Means = -0.8, 95% CI 2-sided [-1.25 to -0.35], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Empagliflozin 25 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1339, ANCOVA; Difference in LS Means = 0.3, 95% CI 2-sided [-0.09 to 0.7], Standard Error of Mean 0.2

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
kilogram (kg) | -2.7 (0.3) | -3.2 (0.3) | -0.5 (0.3)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The change from baseline to Week 26 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and the country as fixed effects, and baseline weight as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -2.25, 95% CI 2-sided [-2.95 to -1.54], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Empagliflozin 25 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1407, ANCOVA; Difference in LS Means = 0.51, 95% CI 2-sided [-0.17 to 1.19], Standard Error of Mean 0.34

6. Secondary Outcome: Change From Baseline in Sitting SBP at Week 12 for All Participants
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
mmHg | -1.7 (0.8) | -2.8 (0.8) | -0.4 (1.0)
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The change from baseline to Week 26 is analyzed using an ANCOVA model using multiple imputations to fill in missing data and is parameterized with treatment groups, randomization strata of HbA1c (≤ 8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No) and the country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.0325, ANCOVA; Difference in LS Means = -2.03, 95% CI 2-sided [-3.89 to -0.17], Standard Error of Mean 0.95
Statistical Analysis 2: Comparison: Sotagliflozin 400 mg vs Empagliflozin 25 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.1565, ANCOVA; Difference in LS Means = 1.1, 95% CI 2-sided [-0.42 to 2.63], Standard Error of Mean 0.78

7. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants. Missing data at Week 26 were assigned a status of nonresponder in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
percentage of participants | 12.1 | 11.7 | 3.9
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; The percentage difference between treatment groups using the Cochran-Mantel-Haenszel test stratified by the randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), and the randomization strata of mean SBP (<130, ≥130 mmHg) at the screening; Test type: Superiority; p = 0.0048, Cochran-Mantel-Haenszel; percentage difference = 8.1, 95% CI 2-sided [3.36 to 12.89]

8. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26
Time Frame: Week 26
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
Number analyzed (Participants) | 307 | 309 | 154
percentage of participants | 32.6 | 35.6 | 15.6
Statistical Analysis 1: Comparison: Sotagliflozin 400 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Percentage Difference = 16.9, 95% CI 2-sided [9.26 to 24.52]

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to 26 weeks) + 4 weeks (Approximately 30 weeks)
Description: Safety population included all randomized participants who received at least one dose of study drug.
Groups:
- Sotagliflozin 400 mg: Following a 2-week run-in period, sotagliflozin 400 mg (milligrams) administered as two 200 mg tablets and one placebo capsule (identical to empagliflozin capsule in appearance), once daily before the first meal of the day for up to 26 weeks.
Arm/Group | Sotagliflozin 400 mg | Empagliflozin 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/307 | 1/309 | 0/154
Serious Adverse Events (participants affected / at risk) | 10/307 | 13/309 | 9/154
Other Adverse Events (participants affected / at risk) | 58/307 | 68/309 | 39/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotagliflozin 400 mg (N=307) | Empagliflozin 25 mg (N=309) | Placebo (N=154)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sotagliflozin 400 mg (N=307) | Empagliflozin 25 mg (N=309) | Placebo (N=154)
Headache (Nervous system disorders) | 7 | 8 | 6
Constipation (Gastrointestinal disorders) | 3 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 10 | 8 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 6 | 9
Any Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 9 | 7
Documented Symptomatic Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 8 | 3
Genital infection fungal (Infections and infestations) | 7 | 5 | 0
Influenza (Infections and infestations) | 5 | 9 | 5
Nasopharyngitis (Infections and infestations) | 12 | 20 | 5
Urinary tract infection (Infections and infestations) | 11 | 8 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 5 | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03351478/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03351478/SAP_001.pdf